CLINICAL TRIAL: NCT03455244
Title: Angiogram Based Fractional Flow Reserve in Patients With Multi-Vessel Disease
Status: Completed | Type: Observational
Sponsor: CathWorks Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CWX-04
Record Dates: First submitted 2018-02-28; First posted 2018-03-06 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Multi Vessel Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: FFRangio — FFRangio is a non-invasive image-based software device that provides physicians with a quantitative analysis of functional significance of the coronary lesion, similar to invasive FFR (Fractional Flow Reserve), and a qualitative three-dimensional model of the demonstrated coronary arteries, during routine PCI procedure. The CathWorks FFRangio software device is able to perform all required processing and calculations, based only on angiography images and hemodynamics information that are acquired during the coronary catheterization procedure.
  The CathWorks FFRangioTM technology does not require any additional use of invasive devices, or any additional vasodilation treatment, as required by other known FFR techniques.

SUMMARY:
This is a prospective, observational, single-center, single-arm, clinical trial designed to assess the efficacy of FFRangio in measuring FFR obtained from angiography compared to Invasive FFR for diagnosing hemodynamically significant coronary stenosis in Multi-Vessel Disease.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age.
* Patients with stable angina or unstable angina or NSTEMI, with at least 1 stenoses ≥ 50% in two main vessels (LAD, LCX and/or RCA) each and in whom invasive FFR is being assessed at these stenoses.
* Patients undergoing invasive FFR with Adenosine, ATP or Papaverine used as hyperemic stimulus.
* Written, informed consent.

Exclusion Criteria:

* Contraindication for FFR examination or administration of vasodilators.
* Clinical presentation of an acute infarct (STEMI) or presented with STEMI in past year.
* CTO in a target vessel.
* Prior CABG, valvular surgery, TAVI/TAVR, or heart transplantation.
* Known LVEF ≤45%.
* Arteries supplying akinetic or severe hypokinetic territories if already known based on prior imaging.
* TIMI Grade 2 or lower at baseline.
* Target lesions involve Left Main (stenosis ≥50%.)
* In-stent restenosis in a target vessel.
* Heavily diffused atherosclerosis diseases defined as the presence of diffuse, serial gross luminal irregularities present in the majority of the coronary tree.
* Target coronary vessels are supplied by major collaterals.
* Lesion is in ectatic segment which includes dilatation in diameter at least 1.5 times that of the adjacent normal coronary artery.
* Coronary angiograms not acquired per instructions as defined in the Study Protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with stable angina, unstable angina or NSTEMI who are referred to coronary angiography, have multi-vessel coronary artery disease and have an invasive FFR measurement at two lesions at minimum. Each subject will undergo both the standard invasive FFRs and the investigational FFRangio.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of the dichotomously scored FFRangio measured index compared to invasive FFR | 1 hour
  Sensitivity and specificity of the dichotomously scored FFRangio measured index per vessel as compared with invasively-derived FFR; Index ≤ 0.80 is scored "positive" while Index > 0.8 is negative.

SECONDARY OUTCOMES:
Continuously scored FFR (FFRangio and Invasive FFR). | 1 hour
  Regression of FFRangio on continuous FFR, with slope, intercept and the correlation coefficient.
Accuracy, Positive predictive value and negative predictive value per vessel and per lesion | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Gifu Heart Center, Gifu, Japan

IPD SHARING:
Plan to Share IPD: No